CLINICAL TRIAL: NCT03562286
Title: Open Spina Bifida Fetoscopic Repair Project
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medicina Perinatal Alta Especialidad, México (Other)
Collaborators: Universidad de Monterrey (Other)
Responsible Party: Principal Investigator, Gerardo Sepúlveda González, Fetal Surgery Coordinator Hospital Christus Muguerza Alta Especialidad, Medicina Perinatal Alta Especialidad, México
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Estudio No.414
Record Dates: First submitted 2018-02-13; First posted 2018-06-19 (Actual); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Myelomeningocele
Keywords: Open spina bifida; spinal dysraphism
MeSH Terms: conditions — Meningomyelocele; Spina Bifida Cystica; Spinal Dysraphism | interventions — Fetoscopy

STUDY DESIGN:
Intervention Model Description: Intervention model: single group assignment Masking: None (Open label) Primary purpose: treatment
Masking Description: Open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Fetoscopy (Experimental): All participants will undergo fetoscopic repair of open spina bifida
  Interventions: Procedure: Fetoscopy

INTERVENTIONS:
Procedure: Fetoscopy — Performing a minimally invasive procedure using a fetoscopic technique in order to access to amniotic cavity and make the endoscopic repair of the fetal neural tube defect.
  Other Names: Fetal surgery

SUMMARY:
The aim of the study is to assess a new fetal surgery approach to repair open spina bifida. The fetal group hypothesis is to perform a minimally invasive procedure using a fetoscopic technique in order to access to amniotic cavity and make the endoscopic repair. This approach will allow investigators to make the closure of the defect and avoid the use of an hysterotomy, reducing the risk of maternal complications as uterine dehiscence (rupture), hemorrhage and preterm premature rupture of membranes (PPROM), the patient also will be able to have a vaginal delivery.

DETAILED DESCRIPTION:
Spina bifida can be a devastating neurological congenital anomaly . It results from incomplete middleline closure of the neural tube between 22 and 28 embryological days. Its incidence is approximately 1 per 1,000 / 2,000 births. It is considered the most common congenital anomaly of the central nervous system that is compatible with life, 90% of the defects are lumbar and sacral.

1. The most frequent form is myelomeningocele (MMC), characterized by the extrusion of the spinal cord into a sac filled with cerebrospinal fluid (CSF), and is associated with lower limb paralysis and bowel and bladder neurological dysfunction.
2. The majority of MMCs can be diagnosed between before 20 weeks. MMC is associated with Chiari II malformation, which includes a constellation of anomalies such as hindbrain herniation, brainstem abnormalities, low-lying venous sinuses and a small posterior fossa.The Chiari II malformation can have deleterious effects on motor, cranial nerve and cognitive functions. Postnatally most MMC patients develop hydrocephalus and require a ventriculoperitoneal shunt. Shunts require lifelong monitoring and have a high failure rate due to infection, obstruction, and fracture.

Experimental studies using animal models have shown that prenatal coverage of a spina bifida-like lesion can preserve neurological function and reduce or reverse hindbrain herniation.These studies suggest a "two-hit" hypothesis in which the ultimate neurologic deficit results from a combination of the failure of normal neural-tube closure (first hit) with secondary spinal cord injury resulting from prolonged exposure of sensitive neural elements to the amniotic fluid (second hit mechanism).

Based on this hypothesis, open fetal surgical repair of MMC was proposed, and the recent publication of the NICHD sponsored randomized controlled trial demonstrated clear neonatal benefit of open in-utero fetal surgical repair of MMC. The study showed a reduction in the incidence of hydrocephalus and in the radiographic severity of hindbrain herniation (relative risk: 0.67; 95% confidence interval: 0.56-0.81).

Open in-utero fetal surgery is not without risk and the NICHD study (MOMS Trial) showed an elevation in maternal-fetal morbidity/risk when compared to the postnatally treated group, including higher risk for chorioamniotic separation (26% vs. 0%, respectively), maternal pulmonary edema (6% vs. 0%), oligohydramnios (21% vs. 0%), placental abruption (6% vs. 0%), spontaneous membrane rupture (46%; RR: 6.15; 95% CI: 2.75-13.78), spontaneous labor (38%; RR: 2.80, 95%CI: 1.51-5.18), maternal blood transfusion (9%; RR: 7.18; 95%CI: 0.90-57.01), and preterm delivery before 34 weeks (46%; RR: 9.2; 95%CI: 3.81-22.19). The reason for the increased incidence of these complications is related to the nature of the open fetal procedure, which involves a multi-faceted invasive approach including maternal laparotomy, large hysterotomy with uterine edge stapling, and open fetal repair of the spina bifida defect that may involve manipulation and exposure of the fetus for a significant amount of time.

Fetal endoscopic surgery has progressed rapidly over the past decades and the investigators are now able to perform a number of intricate procedures inside the uterus with specially designed instruments. These procedures include laser therapy for Twin-twin-transfusion syndrome, fetal cystoscopy and fulguration of posterior urethral valves, release of amniotic bands, and placement of various shunts and balloons inside fetal structures and cavities (peritoneal, pleural, cardiac, and trachea).

Fetoscopy offers a less invasive therapeutic option that could reduce a number of the morbidities (both maternal and fetal) related to open fetal procedures.

A few animal studies and some clinical human experience with fetoscopic repair of MMC have been reported showing the feasibility of covering the defect with a patch and sealant, or even in performing a full repair. These repairs have been accomplished using at least two (and sometimes more) entry ports through the uterine wall. Kohl et al. in Germany, have demonstrated the feasibility of performing a complete percutaneous fetoscopic repair of MMC using carbon dioxide to distend the uterus and provide a dry working area for the surgeon to perform the repair.

These investigators described a two-layer covering technique using an absorbable patch (Durasis, Cook, Germany) and sutures. However, while they showed that the procedure is feasible, their percutaneous technique with complete two layer surgical closure of the defect using sutures was associated with prolonged operative time and significant maternal and obstetrical morbidities.

Fetoscopy in a CO2 gas filled uterus has been recently reported by groups in Bonn, Germany (Kohl et al) and Sao Paulo, Brazil (Pedreira et al). The fetoscopic technique the investigators use has been developed and tested in a fetal sheep model of MMC by the investigators group and others (Peiro et al). This fetoscopy technique has now been employed by a group of investigators, in human fetal surgery cases in Houston, Texas, Monterrey México and in Shiraz, Iran showing its feasibility and applicability to the human uterus and fetus, and demonstrating an improved degree of flexibility in terms of access to the fetus regardless of placental location. The technique is designed to decrease the maternal risks of open uterus fetal surgery while maintaining a similar level of fetal benefit as seen in the MOMS trial.

The investigators technique employs general deep anesthesia and an open abdomen/exteriorized (but closed) uterus methodology that allows the minimally invasive closure of the fetal neural tube using the same closed skin repair currently employed at another US centers using the open uterus approach. The technique employs a novel approach to low pressure uterine distention using the same carbon dioxide gas 8-12 mmHg that others attempting fetoscopic repair have used, but employing a much lower gas flow rate and pressure. In addition, this technique allows a significantly quicker neural tube repair because of improved access to the fetus, ability to manipulate the fetus into the required position, and superior port placement resulting from the exteriorized maternal uterus.

The technique consist in a three access ports (10 French each) and these can be sutured into the uterus allowing a closed seal and minimizing gas leakage. Finally, a 2-3 mm Storz surgical sets enables a full surgical repair to be performed via a fetoscopic approach.

There have been reports about sheep model, with dual access port fetoscopic neural tube closure using a 12 french cannula, a second 9 french cannula, a cover patch, and a medical sealant with similar results to that seen with open fetal surgical repair in the same sheep model. Using the knowledge and expertise gained with more than 3 years of experience in fetoscopic sheep surgery, Dr. Peiro has now performed 8 minimally invasive repairs on human patients in Barcelona (Vall D'Hebron Hospital, Instituto Nacional de Perinatologia, Mexico City, Mexico). Also there have been reports at Texas Childrens Hospital ( Belfort) using two ports technique in order to successfully repair the defect.

The neurosurgical repair proposed in this protocol will involves release of the placode, dissection of the surrounding skin and attempted primary closure of the defect using available skin. In those cases where the investigators are able to complete the procedure with full skin closure of the defect, the only difference between the open uterus procedure and the fetoscopic procedure, will be that the surgery will be done fetoscopically rather than through an open uterine incision. If the investigator group is unable to close the skin primarily despite best fetoscopic efforts, the option of performing/completing the repair as an open procedure exists and will be offered to the patient previous counselling of the maternal morbidity. The patient is monitored in hospital until ready for discharge.

Approximately 6 weeks after the surgery a post-procedure fetal MRI will be performed. If there is evidence of good closure of the neural tube defect and reversal of the Chiari II malformation, a vaginal delivery can be attempted based on obstetric criteria. Patients will be followed in person every 3-4 months after birth to 12 months at the Spina Bifida Clinic at Christus Muguerza Alta Especialidad. Remaining visits will be yearly up to 5 years. If this is not possible, questionnaire(s) will be mailed to the participants and records will be requested from the treating neurosurgeon on this same schedule.

ELIGIBILITY:
Inclusion Criteria:

1. - Pregnant women - maternal age 18 years old or older and capable of consenting for their own participation in the study
2. - Singleton pregnancy
3. - Myelomeningocele with the upper boundary located between T1 and S1
4. - Evidence of hindbrain herniation (confirmed on MRI) to have Arnold Chiari type II malformation)
5. - Absence of chromosomal abnormalities and associated anomalies.
6. - Gestational age at the time of the procedure will be between 19 to 26 weeks
7. - Normal karyotype and / or normal chromosomal microarray (CMA) by invasive testing (amniocentesis or CVS). If there is a balanced translocation with normal CMA with no other anomalies the candidate can be included. Patients declining invasive testing will be excluded.

Exclusion Criteria:

1. - Fetal anomaly unrelated to myelomeningocele
2. - Sever kyphosis
3. - Increased risk for preterm labor included short cervical length (<15 mm), history of incompetent cervix with or without cerclage, and previous preterm birth
4. - Placental abnormalities (previa, abruption, accreta) known at time of enrollment
5. - A prepregnancy body mass index > or equal to 35 Kg/m2
6. - Contraindications to surgery including previous hysterotomy (whether from a previous classical cesarean, uterine anomaly such as an arcuate or bicornuate uterus, mayor myomectomy resection or previous fetal surgery) in active uterine segment.
7. - Technical limitations precluding fetoscopic surgery, such as uterine fibroids, fetal membrane separation, and uterine anomalies.
8. - Maternal fetal Rh isoimmunization, Kell sensitization or neonatal alloimmune thrombocytopenia affecting the current pregnancy
9. - Maternal HIV, Hepatitis B/C status positive
10. - Maternal medical condition that is a contraindication to surgery or anesthesia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women with singleton pregnancy and fetus with myelomeningocele with the upper boundary located between T1 and S1
Enrollment: 45 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Capability to achieve successful closure of the myelomeningocele by fetoscopic surgery | Time of procedure (day 0)
  Binary variable (yes/no) describing if the neural tube defect (myelomeningocele) has been successfully closed (placed dissected and dropped into the open spinal canal, cystic tissue resected and edges closed to the midline), by fetoscopic surgery, and without conversion to open surgery.

SECONDARY OUTCOMES:
Surgery time (minutes) | Time of procedure in minutes (day of surgery / day 0)
  Time between the skin incision and skin closure
Delivery gestational age (weeks and days) | From surgery and up to 21 weeks after the procedure
  Gestational age at birth
Premature rupture of membranes PROM (weeks and days) | Between the surgery to 37 weeks of pregnancy (18 weeks after repair)
  Amniotic fluid leakage before onset of labor
Chorioamnionitis | Between the surgery and delivery (up to 20 weeks after repair)
  The presence or absence of an intrauterine infection
Mode of delivery | Delivery, up to 21 weeks after surgery
  Vaginal or cesarean delivery
Neurodevelopment evaluation by Bayley Scales of infant development II | Up to 24 months after birth
  Score of the Mental Developmental Index of the Bayley Scales of Infant Development II at 24 months of age. The score ranges from 50 (minimum) to 150 (maximum). A score of <70 indicates severe developmental delay; 70-84 indicates moderate delay; >85 indicates no delay.
Childhood motor function on physical examination | 24 months after birth
  Difference between the anatomic upper border of the lesion level and motor function based on the physical examination at 24 months of age. A positive score of 2 indicates a functional level 2 vertebrae higher than lesion level. A score of -2 indicates a function level 2 vertebrae lower than the lesion level.
Ventriculoperitoneal shunt | After birth and up to 12 months
  Need for a cerebrospinal fluid shunt within the first year of life

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Christus Muguerza Alta Especialidad, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: No